CLINICAL TRIAL: NCT03471507
Title: Efficacy of a Topical Pain Relief Spray Containing Herbal Oil Extracts (Bonipar) Among Individuals With Acute and Chronic Musculoskeletal Pain
Brief Title: Bonipar for Acute and Chronic Musculoskeletal Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Winston Parris, MD (Other)
Responsible Party: Sponsor-Investigator, Winston Parris, MD, Professor Emeritus, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00081546
Record Dates: First submitted 2018-03-14; First posted 2018-03-20 (Actual); Results first posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-08

CONDITIONS: Chronic Pain; Musculoskeletal Pain
MeSH Terms: conditions — Chronic Pain; Musculoskeletal Pain

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to one of two study groups (Bonipar or diclofenac topical solution 1.5%), utilizing a predetermined randomization schedule in a 1:1 ratio.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The bottles will be labelled by pharmacy either "Drug A" or Drug B" according to their designation with a label affixed to cover any drug manufacturing labeling. Only the dispensing pharmacy will not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bonipar (Experimental)
  Interventions: Drug: Bonipar
- Diclofenac topical solution 1.5% (Active Comparator)
  Interventions: Drug: Diclofenac sodium topical solution 1.5%

INTERVENTIONS:
Drug: Bonipar — Apply 2 pumps 2 times a day to be applied topically on the affected area during a two week treatment period.
  Arms: Bonipar
Drug: Diclofenac sodium topical solution 1.5% — Apply 2 pumps 2 times a day to be applied topically on the affected area during a two week treatment period.
  Arms: Diclofenac topical solution 1.5%

SUMMARY:
This study is a non-inferiority study comparing efficacy and onset of action between the herbal extracts topical solution, Bonipar, and diclofenac sodium topical solution, diclofenac topical solution 1.5%.

DETAILED DESCRIPTION:
This study is a non-inferiority study comparing efficacy and onset of action between the herbal extracts topical solution, Bonipar, and diclofenac sodium topical solution, diclofenac topical solution 1.5% (approved by the FDA as a topical analgesic). Approximately 168 Duke patients will be recruited from Duke Pain Clinic, and selected Duke primary care practices. Individuals who report acute (less than 3 months duration) or chronic musculoskeletal pain of any intensity will be considered for enrollment into the study. After obtaining consent, eligible subjects will be will be randomized to receive Bonipar or diclofenac topical solution 1.5%.

ELIGIBILITY:
INCLUSIONARY CRITERIA:

* Subject with acute and chronic localized musculoskeletal pain
* Ages 18 to 80 years
* Subjects of all races, gender or ethnic groups
* Female subjects of childbearing age must have a negative pregnancy test Female subjects of childbearing age who are sexually active must agree to use appropriate contraceptive measures for the duration of the study. Medically acceptable contraceptives include: (1) surgical sterilization (such as tubal ligation or hysterectomy), (2) approved hormonal contraceptives (such as birth control pills, patches, implants or injections), (3) barrier methods (such as a condom or diaphragm) used with a spermicide, or (4) an intrauterine device (IUD).
* Willing to provide written informed consent
* Patients taking opioid or NSAID for their musculoskeletal pain may be included if pain is inadequately controlled

EXCLUSIONARY CRITERIA:

* Patients meeting any of the following criteria will be excluded from the study: Use within 3 days of any topical agents on the affected area
* Subject with active skin lesions or skin disease or with cutaneous manifestations of systemic illnesses
* Subject with history of uncontrolled diabetes (A1C of more than 9)
* Subject with history of uncontrolled hypertension (SBP > 160 and DBP > 95)
* Subject with active uncontrolled GERD (defined as more than 2 episodes per week) or history of peptic ulcer disease
* Subject with active cancer, spinal cord lesions or spine surgery
* Subject with allergies to diclofenac or to other non-steroid anti-inflammatory drugs (NSAID)
* Known allergies to any oils, methyl salicylate and/or camphor
* Subject is pregnant or lactating
* Subject with history of heart attack, stroke or blood clot, or recent coronary artery bypass graft surgery (CABG) (i.e., within the last six months)
* Subject with history of alcohol or drug abuse within 1 year
* Subject with history of severe cardiac, liver or kidney disease or any other medical condition that may interfere with the subject's ability to participate in the study as determined by the Investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2022-09-22 (Actual); Study Completion 2022-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lance Roy, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bonipar | Diclofenac Topical Solution 1.5%
Started | 81 | 83
Completed | 78 | 78
Not Completed | 3 | 5
Not completed — Lost to Follow-up | 1 | 3
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bonipar | Diclofenac Topical Solution 1.5% | Total
Number analyzed (Participants) | 81 | 83 | 164
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (16.6) | 54.2 (15.1) | 52.8 (15.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 52 | 99
  Male | 34 | 31 | 65
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 74 | 75 | 149
  Unknown or Not Reported | 3 | 4 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 10 | 16
  White | 65 | 65 | 130
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 4 | 5 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 81 | 83 | 164

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain as Measured by Subjective Pain Intensity Rating (SPIR)
Description: The SPIR is a patient-reported graduated scale where 0 = no pain and 10 = the maximum pain imaginable.
Time Frame: Baseline (approximately 24 hours before consent) to approximately 1 week post administration of study drug (or comparator)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bonipar | Diclofenac Topical Solution 1.5%
Number analyzed (Participants) | 81 | 83
score on a scale | -2.3 (2.0) | -2.6 (1.9)
Statistical Analysis 1: Comparison: Bonipar vs Diclofenac Topical Solution 1.5%; Test type: Other; p = 0.46, Regression, Linear; Adjusted for age and sex

2. Secondary Outcome: Number of Participants Who Experienced Adverse Effects and/or Complications
Time Frame: Up to approximately 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Bonipar | Diclofenac Topical Solution 1.5%
Number analyzed (Participants) | 81 | 83
Participants | 18 | 21

3. Other Pre Specified Outcome: Time to the Onset of Action (the First Feeling of 20% Pain Reduction)
Description: Time to the onset of action measured in minutes.
Time Frame: Up to 1 hour
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Bonipar | Diclofenac Topical Solution 1.5%
Number analyzed (Participants) | 81 | 83
minutes | 21 [15 to 45] | 30 [15 to 45]

ADVERSE EVENTS:
Time Frame: Up to approximately 1 week
Arm/Group | Bonipar | Diclofenac Topical Solution 1.5%
All-Cause Mortality (participants affected / at risk) | 0/81 | 0/83
Serious Adverse Events (participants affected / at risk) | 0/81 | 0/83
Other Adverse Events (participants affected / at risk) | 18/81 | 21/83
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bonipar (N=81) | Diclofenac Topical Solution 1.5% (N=83)
Change in blood pressure (Cardiac disorders) | 1 | 0
Dizziness and increased heart rate (Cardiac disorders) | 1 | 0
Mild tinnitus (Ear and labyrinth disorders) | 1 | 0
Eye irritation (Eye disorders) | 1 | 0
Diarrhea with blood in the stool (Gastrointestinal disorders) | 1 | 0
GI discomfort (Gastrointestinal disorders) | 0 | 1
Dysgeusia (General disorders) | 1 | 0
Epistaxis (General disorders) | 0 | 1
Head Congestion (General disorders) | 1 | 0
Headache (General disorders) | 1 | 1
Increase in leg (calf and thigh) pain (General disorders) | 0 | 1
Increase weakness in leg (General disorders) | 0 | 1
Leg Discomfort (General disorders) | 0 | 1
Lump formation in right hand (General disorders) | 0 | 1
Lump formation on left thumb (General disorders) | 1 | 0
Metallic taste (General disorders) | 1 | 1
Migraine (General disorders) | 0 | 1
Nasal Congestion (General disorders) | 1 | 0
Neck pain (General disorders) | 1 | 0
Radiating shoulder pain (General disorders) | 1 | 0
Rhinorrhea (General disorders) | 1 | 1
Right upper eyelid twitch (General disorders) | 0 | 1
Sneezing (General disorders) | 1 | 0
Treatment site swollen (General disorders) | 0 | 1
Abdominal Muscle Spasm (Musculoskeletal and connective tissue disorders) | 1 | 0
Altered Gait (Nervous system disorders) | 1 | 0
Dysesthesia (Nervous system disorders) | 1 | 1
Dysesthesia/Numbness (Nervous system disorders) | 1 | 1
Numbness (Nervous system disorders) | 0 | 1
Tingling in foot and calf of treated leg (Nervous system disorders) | 0 | 1
Tingling in left hand (Nervous system disorders) | 1 | 0
Tingling toes in treated ankle (Nervous system disorders) | 1 | 0
Vivid Dreams (Psychiatric disorders) | 0 | 1
Allergies (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough/congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dryness (Skin and subcutaneous tissue disorders) | 0 | 1
Dryness around freckle (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Itching (Skin and subcutaneous tissue disorders) | 0 | 4
Mild skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritic Palms (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Rash on both sides of neck (Skin and subcutaneous tissue disorders) | 1 | 0
Redness (Skin and subcutaneous tissue disorders) | 0 | 1
Redness along wrist (Skin and subcutaneous tissue disorders) | 0 | 1
Redness on shoulder (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-01): https://cdn.clinicaltrials.gov/large-docs/07/NCT03471507/Prot_SAP_000.pdf